CLINICAL TRIAL: NCT07345637
Title: A Single-Arm, Open-Label, Dose-Escalation and Expansion Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of FXS887 in Patients With Advanced Solid Tumors
Brief Title: Phase I Study of FXS887 in the Treatment of Solid Tumors
Acronym: FXS887-I101
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FXS887-I101
Record Dates: First submitted 2025-12-23; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor Refractory to Conventional Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FXS887 (Experimental): This is a single-arm, open-label, dose-escalation and dose-expansion Phase I clinical trial evaluating the safety, tolerability, pharmacokinetics, and preliminary efficacy of FXS887 in patients with advanced solid tumors. It mainly consists of two parts: the Phase Ia dose-escalation study and the Phase Ib dose-expansion study. Participants will receive FXS887 orally once-daily at determined dose levels on a 28-day cycle.
  Interventions: Drug: FXS887

INTERVENTIONS:
Drug: FXS887 — FXS887 is an innovative ATR inhibitor targeting ATR kinase.

SUMMARY:
This is a single-arm, open-label, dose-escalation and dose-expansion Phase I clinical trial evaluating the safety, tolerability, pharmacokinetics, and preliminary efficacy of FXS887 in patients with advanced solid tumors. FXS887 is a innovative ATR inhibitors of a class of small-molecule inhibitors targeting ATR kinase.

DETAILED DESCRIPTION:
There will be two parts for this study:

Phase 1a is a dose-escalation, open-label study designed to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of FXS887 in patients with advanced solid tumors. Approximately 14 subjects are expected to be enrolled.

Dose escalation will adopt a combination of "accelerated titration" and "3+3" design. The initial 2 dose cohorts will use the accelerated titration, while the 3+3 design will be implemented starting in other dose cohorts. If a Dose Limiting Toxicity (DLT) event or a study treatment-related adverse event of grade ≥2 occurs during the DLT observation period, the current dose cohort will switch to the 3+3 design. Eligible subjects will receive oral FXS887 once daily. The DLT observation period is within 28 days after the first dose (Cycle 1), followed by multiple-dose studies in Cycle 2 and subsequent cycles. Treatment will continue until the subject experiences disease progression, death, unacceptable toxicity, withdrawal of informed consent, or other reasons requiring discontinuation of study treatment (whichever occurs first).

Phase 1b is an open-label, dose-expansion study that plans to enroll eligible patients with advanced solid tumors. The sample size will be determined based on the results of the Phase 1a, to further evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of FXS887 at the recommended expansion dose(s).

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years, male or female;
2. Participants must fully understand the requirements of the study and voluntarily sign the written informed consent;
3. Participants with histologically/cytologically confirmed advanced solid tumors who have received ≥ 1 line of systemic therapy prior to enrollment in the study and experienced failure of standard therapy (disease progression or intolerance);
4. Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, participants must have at least one measurable target lesion;
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1;
6. Estimated life expectancy of ≥ 12 weeks;
7. Participants must have adequate organ and bone marrow function.
8. For female participants of childbearing age, the serum pregnancy test within 7 days prior to the first dose of the study drug must be negative; eligible participants of reproductive potential (both males and females) must agree to use reliable contraceptive methods (hormonal, barrier, abstinence, etc.) with their partners during the study period and for at least 6 months after the last dose of the study drug.

Exclusion Criteria:

1. Within the washout period of prior anti-tumor medication treatment (4 weeks or 5 half-lives after the last dose, whichever is longer) prior to the first dose of FXS887;
2. Have participated in another clinical study within 4 weeks prior to the first dose of FXS887;
3. Have a history of hypersensitivity to any known components of FXS887 or its analogues;
4. Have intolerance to ATR inhibitors or have received ATR inhibitors within 4 weeks or 5 half-lives (whichever is longer) prior to the first dose of FXS887;
5. Need to take strong CYP3A inhibitors and/or inducers, as well as P-gp (P-glycoprotein) inhibitors and/or inducers within 14 days (or 5 half-lives, whichever is longer) prior to the first dose of FXS887 and during the study period;
6. Need to take drugs known to prolong the QTc interval during the study period;
7. Have had other malignant tumors within 2 years prior to the first dose of FXS887, except for local tumors that have been cured and judged by the investigator to have a low risk of recurrence;
8. Have received radiation therapy within 14 days prior to the first dose of FXS887;
9. Have not recovered from adverse events caused by prior anti-cancer treatment (recovered to Grade 1 or baseline), except for alopecia, pigmentation of any grade, Grade ≤2 peripheral sensory neuropathy, and items explicitly specified in the inclusion criteria;
10. Have refractory nausea and vomiting, chronic gastrointestinal diseases including but not limited to active diverticulitis and symptomatic peptic ulcers, inability to swallow oral medications, or a history of extensive small bowel resection or other conditions that significantly impair gastrointestinal absorption as judged by the investigator;
11. Have undergone major surgery within 2 weeks prior to the first dose or have not recovered from surgical complications;
12. Have primary central nervous system (CNS) tumors, meningeal metastasis, spinal cord compression, or brainstem metastasis; participants with known untreated brain metastases or symptomatic or unstable disease are excluded; participants who have completed treatment for brain metastases (radiation therapy or surgery) with stable metastases and no relevant symptoms (without medication control) within 4 weeks prior to the first dose may be enrolled;
13. Have severe cardiovascular diseases;
14. Have uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage and medical intervention;
15. Have active infections requiring treatment (e.g., participants are receiving anti-infective treatment) within 14 days prior to the first dose of FXS887, including Hepatitis C virus (HCV), Human Immunodeficiency Virus (HIV), uncontrolled active Hepatitis B virus (HBV) infection, syphilis infection, known active tuberculosis, etc.
16. Known infection with hepatitis B virus (HBV) or hepatitis C virus (HCV):

    * participants with controlled HBV infection (serum HBV-DNA < 500 IU/mL or < 2,000 copies/mL) are allowed to enroll in this study.
    * participants who are HCV antibody-positive with controlled infection [polymerase chain reaction (PCR) for serum HCV-RNA below the lower limit of detection] are allowed to enroll in this study.
17. History of human immunodeficiency virus (HIV) infection;
18. History of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis requiring steroid therapy, or clinically active ILD;
19. Known substance abuse or psychiatric disorder that may interfere with compliance with study requirements;
20. Participants are pregnant, breastfeeding, or planning to become pregnant during the study period;
21. Investigator considers the participant has other factors that may affect study results or interfere with participation in the entire study, including past or existing medical conditions, treatment or laboratory abnormalities, or unwillingness to comply with study procedures, restrictions, and requirements-any condition deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 14 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-04-28 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with DLTs | Up to Day 28
  DLTs will be assessed during the dose-escalation phase and are defined as toxicities that meet pre-defined DLT criteria and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, intercurrent illness, or concomitant medications that occurs within the first cycle (28 days) of treatment.
Maximum tolerated dose (MTD) or Maximum administered dose(MAD) | Up to 12 Months
  The MTD is defined as the highest dose level at which the proportion of subjects who experience Dose-Limiting Toxicity (DLT) is less than 1/3 during the DLT observation period. If the MTD is not established after the completion of the dose-escalation, the highest safe dose level will be defined as the MAD.
Incidence of Treatment-Emergent Adverse Events (TEAEs)[Safety and Tolerability] | From first dose of study drug until 30 days after the last dose.
  Number and frequency of subjects with adverse events, including changes in vital signs, electrocardiograms (ECGs), physical examinations, and laboratory parameters, graded according to NCI CTCAE v5.0.
Phase 1a: recommended phase 2 dose (RP2D) | Up to 12 Months
  The RP2D (Recommended Phase 2 Dose) determined based on comprehensive consideration of safety, tolerability, PK (pharmacokinetics), PD (pharmacodynamics), and efficacy data.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of FXS887 | From the day of first dose to 30 days after last dose of FXS887
  Maximum observed plasma concentration of FXS887 following single and multiple doses.
Area under the plasma concentration-time curve (AUC)of FXS887 | From the day of first dose to 30 days after last dose of FXS887
  The area under the plasma concentration-time curve of FXS887 following single and multiple doses.
Time to reach maximum plasma concentration (Tmax) of FXS887 | From the day of first dose to 30 days after last dose of FXS887
  Time to reach maximum plasma concentration of FXS887 following single and multiple doses.
Elimination Half-Life (t1/2) of FXS887 | From the day of first dose to 30 days after last dose of FXS887
  Apparent terminal elimination half-life of FXS887 in plasma.
Objective response rate, ORR | From first dose of study drug until the date of first documented disease progression or death from any cause, whichever occurs first, assessed up to 24 months.
  Antitumor activity by evaluation of tumor response assessments based on RECIST 1.1
Progression Free Survival | From first dose of study drug until the date of first documented disease progression or death from any cause, whichever occurs first, assessed up to 24 months.
  Antitumor activity by evaluation of tumor response assessments based on RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No